CLINICAL TRIAL: NCT04049539
Title: Open-Label Phase 2 Trial of Vyxeos in Patients With Intermediate and High-Risk Acute Myeloid Leukemia Who Have Failed an Initial Cycle of Standard Cytarabine and Daunorubicin Chemotherapy
Brief Title: Vyxeos for Re-induction Treatment of Acute Myeloid Leukemia Patients With Persistent Disease After Induction
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Greg Behbehani, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19060; NCI-2019-04724 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Blasts More Than 5 Percent of Bone Marrow Nucleated Cells; Persistent Disease; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (liposome-encapsulated daunorubicin-cytarabine) (Experimental): Within 14-33 days after the start of previous cycle of chemotherapy, patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This phase II trial studies the side effects and how well Vyxeos works in treating patients with intermediate and high-risk acute myeloid leukemia who have failed an initial cycle of standard cytarabine and daunorubicin chemotherapy. Vyxeos is a combination of both chemotherapy drugs cytarabine and daunorubicin contained in a liposome. Drugs used in chemotherapy, such as cytarabine and daunorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cytarabine and daunorubicin given together in liposomes may have fewer side effects and work better than cytarabine and daunorubicin given alone in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the safety and estimate the efficacy of liposome-encapsulated daunorubicin-cytarabine (Vyxeos) in acute myeloid leukemia (AML) patients who have failed to achieve a hypocellular marrow after an initial course of 7+3.

SECONDARY AND/OR EXPLORATORY OBJECTIVES:

I. Determination of rate of morphologic leukemia-free state (MLFS). II. Determination of progression-free survival (PFS), and overall survival (OS) at 2 years.

III. Mass cytometric measurement relative clearance of quiescent leukemia stem/repopulating cells (LSCs) and blasts as compared to the same patient's preceding cycle of 7+3 and to a separate control population receiving re-induction with traditional 7+3.

IIIa. Measurement of blast cell cycle fraction before and after Vyxeos treatment.

IIIb. Relative clearance immunophenotypically abnormal blast and stem cells after Vyxeos.

IIIc. Comparison of efficacy of blast cell and LSC elimination in patients receiving Vyxeos re-induction compared to similar blast cells and LSCs in patients receiving standard 7+3 or 5+2 re-induction.

OUTLINE:

Within 14-33 days after the start of previous cycle of chemotherapy, patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up weekly for 60 days, then at least monthly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject or their legal guardian must be able to provide written informed consent
* Patients must have a diagnosis of acute myeloid leukemia
* Patients must have received standard continuous infusion cytarabine and daunorubicin (cytarabine 100-200 mg/m^2 by continuous infusion on days 1-7 and daunorubicin 45-90 mg/m^2 on days 1-3) within the 14-33 days prior to starting trial treatment and have documented persistent disease (13-29 days from the start of 7+3 treatment). Patients who have received a 7+3 regimen utilizing idarubicin (12 mg/m^2 on days 1-3) in place of daunorubicin may enroll. Persistent disease will be defined as bone marrow cellularity of > 10-20% and bone marrow blast percentage of > 5-10% or clear evidence of immunophenotypically aberrant leukemia cells in the bone marrow. The final determination of persistent AML will be made by the treating physician, but must meet National Comprehensive Cancer Network (NCCN) criteria for persistent disease. Enrollment of patients with less than 20% cellularity or less than 10% blasts will require approval of the principal investigator. Patients who received concomitant treatment with another targeted therapy for AML (e.g. midostaurin) during initial induction may enroll, but will not continue to receive this treatment during Vyxeos treatment
* Patients must be deemed by the treating physician to be unlikely to achieve complete response (CR) without further therapy
* Patients must be deemed by the treating physician to be able to tolerate intensive chemotherapy (similar to 7+3 chemotherapy)
* Normal left ventricular ejection fraction (>= 50% by echocardiography or multi-gated acquisition radionuclide angiocardiography [MUGA]) and lifetime daunorubicin dose of less than 418 mg/m^2 (including recent course of 7+3)
* Eastern Cooperative Oncology Group (ECOG) functional status of 0, 1, or 2
* Aspartate aminotransferase (AST) < 5 x upper limit of normal (ULN) for the local laboratory
* Alanine aminotransferase (ALT) < 5 x ULN for the local laboratory
* Total bilirubin < 1.5 x ULN (except for patients with known Gilbert?s syndrome) for the local laboratory
* Calculated creatinine clearance (according to the Cockcroft-Gault equation) > 40 mL/min OR serum creatinine < 1.5 x the ULN for the local laboratory
* Female patients of childbearing potential must agree to use two forms of contraception from screening visit until 6 months following the last dose of study treatment. Female patients must have a documented negative pregnancy test
* Male patients of childbearing potential having intercourse with females of childbearing potential must agree to abstain from heterosexual intercourse or have their partner use two forms of contraception from screening visit until 90 days until the last dose of study treatment. They must also refrain from sperm donation from screening visit until 90 days following the last dose of study treatment

Exclusion Criteria:

* Acute promyelocytic leukemia (or M3 AML)
* Patients known to have core binding factor AML (defined as presence of t(8;21), inv(16), or other cytogenetically equivalent abnormalities)
* Patients known to have inactivating mutations of TP53 or evidence of an absence of p53 protein activity as indicated by a monosomal karyotype. Monosomal karyotype will be defined as two or more monosomies (loss of an entire chromosome or the entire long arm of a chromosome [such as 7q-]) or a single monosomy in the setting of a complex karyotype. Patients with a complex karyotype without a monosomy are eligible to enroll
* Patients that the treating physician does not feel are able to tolerate intensive chemotherapy
* History of serious (>= grade 3) hypersensitivity reaction to cytarabine, daunorubicin, or any component of the formulation
* Known Wilson's disease or other symptomatic abnormality of copper metabolism (laboratory screening is not required in the absence of clinical or historical evidence of Wilson's disease or other problems of copper metabolism)
* Total lifetime daunorubicin dose of more than 418 mg/m^2 (including recent course of 7+3) or equivalent total doses of other anthracycline medications
* Pregnancy or inability to use highly effective method of contraception for 6 months following last dose of Vyxeos. Potentially fertile patients must have documented negative serum pregnancy test. Breastfeeding should be avoided for at least 14 days after the last dose Vyxeos
* Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control. As infection is a common feature of AML, patients with active infections are permitted to enroll provided that the infection is under control
* Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent and until toxicity from this has resolved to grade 1 or less; if the half-life of the agent is unknown, patients must wait 4 weeks prior to first dose of study treatment. An investigational agent is one for which there is no approved indication by the United States (US) Food and Drug Administration (FDA)
* Patients with psychological, familial, social, or geographic factors that otherwise preclude them from giving informed consent, following the protocol, or potentially hamper compliance with study treatment and follow-up
* Any other significant medical condition, including psychiatric illness or laboratory abnormality, that would preclude the patient participating in the trial or would confound the interpretation of the results of the trial
* Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Other malignancy currently requiring active therapy (except minor surgery for non-melanoma skin cancer and for hormonal/anti-hormonal treatment, e.g. in prostate or breast cancer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 60 days
  Will be measured by the time to count recovery, incidence of symptomatic cardiac dysfunction, incidence of hepatic or renal toxicity, incidence of severe hemorrhage, and incidence of severe infection. Will be summarized by National Cancer Institute Common Terminology Criteria for Adverse Events version 4, and frequency counts will be tabulated with a focus on severe (grade 3+) adverse events and toxicities that are deemed at least possibly related to study treatment. The incidence of specific toxicities will be calculated as the proportion of patients experience these toxicities over all patients who receive any study drug.
Calculation rate of complete response (CR) and complete response with incomplete hematologic recovery (CRi) | Up to 2 years
  CR and CRi rate will be defined as the proportion of patients who achieve CR or CRi over all evaluable patients. The rates will be provided with 95% binomial confidence intervals.

SECONDARY OUTCOMES:
Progression-free survival | Up to 2 years
  Will be calculated by the method of Kaplan-Meier, with the 2-year estimate provided with 95% confidence interval.
Overall survival | From the date of the first dose of study treatment to death from any cause, up to 2 years
  Will be calculated by the method of Kaplan-Meier, with the 2-year estimate provided with 95% confidence interval.

OTHER OUTCOMES:
Measurement of blast cell cycle fraction | Baseline up to day 42
  Will be exploratory in nature with graphical methods and descriptive statistics provided to gather preliminary information. Nonparametric method such Mann-Whitney U test will be utilized to compare pre and post-treatment data, and box plot or spaghetti plot will be presented to help visualize the trend of change.
Relative clearance immunophenotypically abnormal blast and stem cells | Up to day 42
  Will be exploratory in nature with graphical methods and descriptive statistics provided to gather preliminary information. Nonparametric method such Mann-Whitney U test will be utilized to compare pre and post-treatment data, and box plot or spaghetti plot will be presented to help visualize the trend of change.
Efficacy of blast cell and leukemia stem/repopulating cell (LSC) elimination | Up to day 42
  Will compare the efficacy of blast cell and LSC elimination in patients receiving Vyxeos re-induction compared to similar blast cells and LSCs in patients receiving standard 7+3 or 5+2 re-induction. Will be exploratory in nature with graphical methods and descriptive statistics provided to gather preliminary information. Nonparametric method such Mann-Whitney U test will be utilized to compare pre and post-treatment data, and box plot or spaghetti plot will be presented to help visualize the trend of change.
Number of patients proceeding to stem cell transplantation following Vyxeos treatment | Up to 2 years
  Will be measured and is exploratory in nature. It will be analyzed with descriptive statistics to gather preliminary information and compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory K Behbehani, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu